CLINICAL TRIAL: NCT00003604
Title: A Multi-Center Adjuvant Trial of Outpatient Moderate-Dose Bolus Interleukin-2 for Renal Cancer
Brief Title: Interleukin-2 in Treating Patients With Stage III or Stage IV Kidney Cancer That Has Been Removed With Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Biotherapy Research Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066679; CBRG-9704; NBSG-9704; NCI-V98-1482
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2000-09

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 in treating patients with stage III or stage IV kidney cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the disease free survival and overall survival of patients with resected stage III or IV renal cancer treated with interleukin-2. II. Measure the degree of rebound lymphocytosis generated by this regimen in these patients.

OUTLINE: This is an open label study. Patients receive interleukin-2 IV over 15-30 minutes on 3 consecutive days weekly for 6 weeks, followed by 2 weeks of rest. Patients receive 2 treatment courses, each 8 weeks in duration. Patients are followed every 6 months until death.

PROJECTED ACCRUAL: A total of 20 patients will be accrued within 1 to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV renal cancer that has been completely resected and is at high risk for recurrence, including at least one of the following: Tumor invades adrenal gland or perinephric tissues but not beyond Gerota's fascia (T3a) OR Tumor extending into renal vein, vena cava (T3b) OR Tumor grossly extends into vena cava above diaphragm (T3c) OR Tumor invades beyond Gerota's fascia (T4) OR Any lymph node involvement totally resected (N1-3) OR Completely resected metastases of all sites No brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin less than 3 times upper limit of normal (ULN) AST or ALT less than 3 times ULN Renal: Creatinine no greater than 1.9 mg/dL Cardiovascular: No prior myocardial infarction within 6 months No LVEF less than 35% No primary cardiac arrhythmias beyond occasional PVCs No angina No uncontrolled congestive heart failure No cerebrovascular accident Pulmonary: No dyspnea at rest or requirement for supplemental oxygen Oxygen saturation greater than 90% for patients with symptomatic lung disease Other: Not pregnant or nursing Negative pregnancy test Fetile patients must use effective contraception Temperatures greater than 100.5 degrees F must have occult infection excluded No psychiatric disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent cyclosporine or methotrexate Endocrine therapy: At least 3 weeks since prior corticosteroids No concurrent corticosteroids Radiotherapy: Not specified Surgery: At least 2 weeks since prior surgery Other: At least 3 weeks since prior immunosuppressive medications No concurrent immunosuppressive medications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1997-10

CONTACTS AND LOCATIONS:
Overall Officials: Datchen F. Tai, MD, Study Chair — Cancer Biotherapy Research Group
Locations (3):
- United States (3):
  - Cancer Care Center for Southern Indiana, Bloomington, Indiana
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee